CLINICAL TRIAL: NCT06787144
Title: A Phase 1 Study of ELVN-001 for the Treatment of Chronic Myeloid Leukemia With and Without T315I Mutation in Japanese Participants
Brief Title: ELVN-001 for the Treatment of Chronic Myeloid Leukemia With and Without T315I Mutation in Japanese Participants
Acronym: CML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enliven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELVN-001-105
Record Dates: First submitted 2024-12-16; First posted 2025-01-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: CML (Chronic Myelogenous Leukemia); Chronic Phase CML
Keywords: CML; Tyrosine Kinase Inhibitor; T315I; T315I Mutant; BCR-ABL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1 Dose Escalation (Experimental): ELVN-001 administered in 3+3 dose escalation
  Interventions: Drug: ELVN-001
- Part 2 Dose Exploration (Experimental): ELVN-001 administered to approximately 6 participants per dose level who may be enrolled at or below the dose levels that have been deemed safe and tolerable in Part 1
  Interventions: Drug: ELVN-001

INTERVENTIONS:
Drug: ELVN-001 — Orally once or twice daily

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and determine the recommended dose for further clinical evaluation of ELVN-001 in Japanese patients with chronic phase chronic myeloid leukemia with and without T315I mutations in patients who has failed, or the patient is intolerant to, or not a candidate for, at least 2 prior TKIs.

DETAILED DESCRIPTION:
This first-in-human trial with ELVN-001 is a dose escalation study with the primary purpose to identify the recommended dose(s) for expansion (RDEs) of single agent ELVN-001 in chronic phase CML with or without T315I mutations. The safety, tolerability and pharmacokinetic profile of ELVN-001 will be assessed together with an evaluation of changes in BCR-ABL1 transcript. An understanding of the safety profile, PK and preliminary evidence of anti-CML activity will be used to inform future development of ELVN-001 in adults with CML. By virtue of its predicted pharmacological profile ELVN-001 has the potential to be tolerable and achieve a deep molecular response in patients with CML with or without T315I mutations who have failed, or are intolerant to, or not a candidate for, at least 2 prior TKIs.

ELIGIBILITY:
Inclusion Criteria:

* BCR::ABL1 positive CP-CML that has failed, or the patient is intolerant to, or not a candidate for, at least 2 prior TKIs.
* ECOG performance status of 0 to 2.
* The patient was born in Japan and both parents and grandparents are Japanese.
* Adequate hematologic, hepatic and renal function.
* Prior bone marrow transplant allowed if ≥ 6 months prior to the first dose of ELVN-001.

Exclusion Criteria:

* Treatment with anti-cancer or anti-CML therapy within 7 days or 5 half-lives, whichever is longer.
* History of acute tyrosine kinase inhibitor (TKI)-related pancreatitis within 6 months of study entry. Active chronic pancreatitis, or pancreatic disease due to any cause.
* QTc >470 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of dose limiting toxicities | 28 days
  DLTs will be used to support that the recommended doses for expansion are </= MTD
Part 1: Incidence of adverse events (AEs) | Up to 28 days
  Adverse events will be used to support that the recommended doses for expansion are likely to be tolerable
Part 1: Incidence of clinically significant laboratory abnormalities | Up to 28 days
  Clinically significant laboratory abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable
Part 1: Incidence of clinically significant ECG abnormalities | Up to 28 days
  Clinically significant ECG abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable
Part 2: Incidence of adverse events | Up to 3 years
  Adverse events will be used to support that the dose(s) evaluated in exploration is tolerable
Part 2: Incidence of clinically significant laboratory abnormalities | Up to 3 years
  Clinically significant ECG abnormalities will be used to support that the dose(s) evaluated in exploration is tolerable
Part 2: Incidence of clinically significant ECG abnormalities | Up to 3 years
  Clinically significant ECG abnormalities will be used to support that the recommended dose(s) evaluated in exploration is tolerable

SECONDARY OUTCOMES:
Area under the curve | 6 months
  PK parameter based on measurement of drug concentration in blood over time
Maximum concentration | 6 months
  PK parameter based on measurement of drug concentration in blood
Time of maximum concentration | 6 months
  PK parameter which is the time at which the highest concentration of drug in the blood is measured
Minimum concentration | 6 months
  PK parameter based on the measurement of the drug concentration that is at the lowest level once steady state has been achieved.
Molecular response (MR) | Up to 3 years
  Measured by quantitative polymerase chain reaction of BCR-ABL transcript levels
Duration of Molecular Response | Up to 3 years
  Time from first molecular response (as measured by quantitative polymerase chain reaction of BCR-ABL transcript levels) to loss of response or discontinuation of study drug
Complete Hematologic Response (CHR) | Up to 3 years
  The proportion of patients who achieve a CHR who are not in CHR at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Helen Collins, MD, Study Director — Enliven Therapeutics
Locations (4):
- Japan (4):
  - Akita University Hospital, Akita, Akita
  - Aiiku Hospital, Sapporo, Hokkaido
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No